CLINICAL TRIAL: NCT02593279
Title: AVAD: Asthma With Small Airways Dysfunction. Clinical, Immunobiological, Tomodensitometric Description, Genetic Signature Compared With Asthmatic Population With Proximal Airways Obstruction
Brief Title: AVAD: Asthma With Small Airways Dysfunction
Acronym: AVAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties of enrollment
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL14_0212
Record Dates: First submitted 2015-10-28; First posted 2015-11-02 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: ASTHMA
Keywords: Asthma; phenotype; small; airway; proximal; dysfunction
MeSH Terms: conditions — Asthma; Cerebral Palsy | interventions — Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- asthma with proximal or diffuse lung damage (Active Comparator)
  Interventions: Genetic: asthma with proximal airways obstruction phenotype profile description with clinical, biological, morphologic and genetic elements.
- asthma with small airway prevailing damage (Experimental)
  Interventions: Genetic: asthma with small airways dysfunction phenotype profile description with clinical, biological, morphologic and genetic elements.

INTERVENTIONS:
Genetic: asthma with proximal airways obstruction phenotype profile description with clinical, biological, morphologic and genetic elements. — symptoms, medical history, date of start, date of aggravation, comorbidities, increased factors related to asthma, blood eosinophils, blood periostin, allergologic patch test, igE analysis, tomodensitometric test.
  Arms: asthma with proximal or diffuse lung damage
Genetic: asthma with small airways dysfunction phenotype profile description with clinical, biological, morphologic and genetic elements. — symptoms, medical history, date of start, date of aggravation, comorbidities, increased factors related to asthma, blood eosinophils, blood periostin, allergologic patch test, IgE analysis, tomodensitometric test.
  Arms: asthma with small airway prevailing damage

SUMMARY:
The aim of the study is to describe asthma phenotype with small airways dysfunction, in a multiparametric manner, with clinical, biological, morphological and genetic elements compared with asthma with proximal airways obstruction.

The objective of this study is also to complete the clinical, immunobiological and morphological analysis of asthma with small airways dysfunction.

ELIGIBILITY:
General Inclusion Criteria:

* man or woman
* age ≥ 18 years
* asthma
* inform consent signed
* affiliated to health insurance

Specific inclusion criteria : asthma with proximal airways obstruction GROUP

* Maximal Voluntary Ventilation (MMV)<80%
* MMV / Forced Vital Capacity (FVC)≤70%
* Carbon Monoxide Transfer Coefficient (KcO)>80%

Specific inclusion criteria : asthma with small airways dysfunction GROUP

* Maximal Voluntary Ventilation (MMV)≥80%
* MMV / Vital Capacity(VC)>70%
* Carbon Monoxide Transfer Coefficient (KcO)>80%

General Exclusion Criteria:

* pregnant woman or breastfeeding
* patient participating to other biomedical research
* patient who have participated to other biomedical research within the past 3 months
* patient refusing to sign the inform consent

Specific exclusion criteria :

* Patient who stopped smoking since less than 12 months
* Pathological state related to obstructive distal airway damage
* Broncho-pulmonary infectious disease within the past 4 weeks
* Solid tumor curated by chemotherapy or chest radiotherapy
* Chronic respiratory disease
* Asthma exacerbation within the past 3 months
* Oral or systemic corticotherapy within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
mRNA expression levels. | maximum 4 weeks after the inclusion visit.
  mRNA expression levels will be measured by microarray analysis.

SECONDARY OUTCOMES:
clinical asthma profile : symptoms | maximum 4 weeks after the inclusion visit.
  symptoms
clinical asthma profile : medical history | maximum 4 weeks after the inclusion visit.
  medical history
clinical asthma profile : date of start | maximum 4 weeks after the inclusion visit.
  date of start
clinical asthma profile : date of aggravation | maximum 4 weeks after the inclusion visit.
  date of aggravation
clinical asthma profile : comorbidities | maximum 4 weeks after the inclusion visit.
  comorbidities
clinical asthma profile : increased factors related to asthma. | maximum 4 weeks after the inclusion visit.
  increased factors related to asthma.
biological asthma profile :blood eosinophils | maximum 4 weeks after the inclusion visit.
  blood eosinophils
biological asthma profile : blood periostin | maximum 4 weeks after the inclusion visit.
  blood periostin
biological asthma profile : allergologic patch test | maximum 4 weeks after the inclusion visit.
  allergologic patch test
biological asthma profile : IgE analysis | maximum 4 weeks after the inclusion visit.
  IgE analysis
morphological asthma profile : Chest X Ray (tomodensitometric test). | maximum 4 weeks after the inclusion visit.
  Chest X Ray (tomodensitometric test).

CONTACTS AND LOCATIONS:
Overall Officials: GILLES DEVOUASSOUX, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (4):
- France (4):
  - Cabinets de Pneumologie Liberale, Caluire-et-Cuire
  - Hospices Civils de Lyon, Lyon
  - CABINETS DE PNEUMOLOGIE LIBERALE HIA Desgenettes, Lyon
  - HC pneumo C, Pierre-Bénite